CLINICAL TRIAL: NCT05853588
Title: The Effect Of Toolbox Trainings On Nursing Sensitive Quality Indıcators
Brief Title: The Effect Of Training On Nursing Qualıty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Bircan Kara, PhD Stıdent, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IstanbulUCerrahpaşabkara
Record Dates: First submitted 2023-04-12; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Nurse's Role
Keywords: quality indicators; quality in health; quality in nursing

STUDY DESIGN:
Intervention Model Description: This study in randomized controlled, pretest, posttest and experiment, control group design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): It was determined by lot by the volunteer nurses who accepted to participate in the study.
  Interventions: Other: training
- Control group (No Intervention): It was determined by lot by the volunteer nurses who accepted to participate in the study.

INTERVENTIONS:
Other: training — On-the-job (toolbox) training given to the experimental group and containing brief information, lasting at most 10 minutes
  Arms: Experimental group

SUMMARY:
The aim of this study, in a randomized controlled design with pretest, posttest and control groups, is to determine the effect of on-the-job (toolbox) training given to nurses on nursing-sensitive quality indicators (pain management, pressure sores, patient falls, Peripheral Venous Catheter complications and adverse event reporting). it aims to answer are:

- Does toolbox training have an effect on nursing-sensitive quality indicators? After the training, participants are expected to adapt to quality practices.

This study consists of experimental and control groups. Experimental and control groups were determined by drawing lots with the help of an external expert. Nurses who met the inclusion criteria were included in the lottery.

Inclusion criteria for the experimental and control groups were determined as follows:

* Working in one of the hospital's internal medicine or surgical services
* Having been working in the current service for at least 6 months, apart from past work experience
* Having completed the orientation process to the hospital and taking responsibility for patient care
* Voluntarily agree to participate in the study

DETAILED DESCRIPTION:
This study was carried out to determine the effect of toolbox training on nursing-sensitive quality indicators (pain management, pressure sores, patient falls, peripheral venous catheter complications and adverse event reporting) in a randomized controlled, pre-test, post-test, experimental and control group design.

The population of the study consisted of nurses working in the inpatient services (except the intensive care units) of a training and research hospital in Hatay. A total of 77 nurses working in the experimental and control group services determined by randomization constituted the sample of the research (experimental group: 38 nurses, control group: 39 nurses).

ELIGIBILITY:
Inclusion Criteria:

* Working in one of the hospital's internal medicine or surgical services
* Being working in the current service for at least 6 months apart from past work experience
* Having completed the orientation process to the hospital and taking responsibility for patient care
* To voluntarily agree to participate in the study

Exclusion Criteria:

* Participants who did not meet the inclusion criteria were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Nurse Information Form | before the training
  This form consists of 10 questions in total to determine the demographic study characteristics of the nurses participating in the research.
Nursing Sensitive Quality Indicators Application Information Form (pretest-posttest) | before the training
  Both groups were applied before the on-the-job training to be given to the experimental group and after all trainings were completed. It was prepared in the light of current literature in order to determine the knowledge level of nurses in the experimental and control groups about nursing-sensitive quality indicators and to evaluate the effectiveness of on-the-job training given to the experimental group. A minimum of 0 and a maximum of 100 points can be obtained from this test.
Nursing Sensitive Quality Indicators Implementation Checklists | before the training
  The checklists developed in line with the literature have been developed for the management of pain in the unit, pressure ulcer, risk of falling, Peripheral Venous Catheter complications and adverse event reporting, and consist of five sections.In this test, 1 point is given for each complete application.
Unit Quality Indicators Monitoring Form | before the training
  Data on 5 nursing-sensitive quality indicators (fall rates (in percent), patient rate with correct pain management (as a number), pressure ulcer rates (in percent), Peripheral Venous Catheter complication (as a number) and adverse event reporting rates(in percent) ) followed before and after the training, and data on the average number of hospitalization days are included.

SECONDARY OUTCOMES:
Nursing Sensitive Quality Indicators Application Information Form (pretest-posttest) | At 8 weeks after give all trainings
  Both groups were applied before the on-the-job training to be given to the experimental group and after all trainings were completed. It was prepared in the light of current literature in order to determine the knowledge level of nurses in the experimental and control groups about nursing-sensitive quality indicators and to evaluate the effectiveness of on-the-job training given to the experimental group. A minimum of 0 and a maximum of 100 points can be obtained from this test.
Nursing Sensitive Quality Indicators Implementation Checklists | At 8 weeks after give all trainings
  The checklists developed in line with the literature have been developed for the management of pain in the unit, pressure ulcer, risk of falling, Peripheral Venous Catheter complications and adverse event reporting, and consist of five sections.In this test, 1 point is given for each complete application.
Unit Quality Indicators Monitoring Form | At 8 weeks after give all trainings
  Data on 5 nursing-sensitive quality indicators (fall rates (in percent), patient rate with correct pain management (as a number), pressure ulcer rates (in percent), Peripheral Venous Catheter complication (as a number) and adverse event reporting rates(in percent) ) followed before and after the training, and data on the average number of hospitalization days are included.

OTHER OUTCOMES:
Nursing Sensitive Quality Indicators Implementation Checklists | At the 12th week after all trainings are completed
  The checklists developed in line with the literature have been developed for the management of pain in the unit, pressure ulcer, risk of falling, Peripheral Venous Catheter complications and adverse event reporting, and consist of five sections.In this test, 1 point is given for each complete application.
Unit Quality Indicators Monitoring Form | At the 12th week after all trainings are completed
  Data on 5 nursing-sensitive quality indicators (fall rates (in percent), patient rate with correct pain management (as a number), pressure ulcer rates (in percent), Peripheral Venous Catheter complication (as a number) and adverse event reporting rates(in percent) ) followed before and after the training, and data on the average number of hospitalization days are included.

CONTACTS AND LOCATIONS:
Overall Officials: Betül SÖNMEZ, Ass. prof, Study Director — betul.sonmez@iuc.edu.tr
Locations (1):
- İstanbul Univercity-Cerrahpaşa, Istanbul, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heslop L, Lu S, Xu X. Nursing-sensitive indicators: a concept analysis. J Adv Nurs. 2014 Nov;70(11):2469-82. doi: 10.1111/jan.12503. Epub 2014 Aug 12. PMID 25113388
- [Result] Driscoll A, Grant MJ, Carroll D, Dalton S, Deaton C, Jones I, Lehwaldt D, McKee G, Munyombwe T, Astin F. The effect of nurse-to-patient ratios on nurse-sensitive patient outcomes in acute specialist units: a systematic review and meta-analysis. Eur J Cardiovasc Nurs. 2018 Jan;17(1):6-22. doi: 10.1177/1474515117721561. Epub 2017 Jul 18. PMID 28718658
- [Result] Donabedian A. The quality of care. How can it be assessed? JAMA. 1988 Sep 23-30;260(12):1743-8. doi: 10.1001/jama.260.12.1743. PMID 3045356
- [Result] Cavazza, N. & Serpe, A. 2010, The Impact of Safety Training Programs on Workers' Psychosocial Orientation and Behaviour. Revue internationale de psychologie sociale, 23, 187-210.
- [Result] Amiri M, Khademian Z, Nikandish R. The effect of nurse empowerment educational program on patient safety culture: a randomized controlled trial. BMC Med Educ. 2018 Jul 3;18(1):158. doi: 10.1186/s12909-018-1255-6. PMID 29970054
- [Result] Burke MJ, Sarpy SA, Smith-Crowe K, Chan-Serafin S, Salvador RO, Islam G. Relative effectiveness of worker safety and health training methods. Am J Public Health. 2006 Feb;96(2):315-24. doi: 10.2105/AJPH.2004.059840. Epub 2005 Dec 27. PMID 16380566
- [Derived] Kara B, Sonmez B. The Effect of Toolbox Trainings on Nursing Sensitive Quality Indicators: A Randomized Controlled Trial. J Nurs Scholarsh. 2025 May;57(3):439-451. doi: 10.1111/jnu.13051. Epub 2025 Jan 31. PMID 39888187